CLINICAL TRIAL: NCT03695965
Title: Magnetic Resonance Imaging Evaluation of Lateral Ankle Instability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: MRILAI
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients with history of ankle trauma or chronic lateral ankle pain
  Interventions: Procedure: magnetic resonance imaging.

INTERVENTIONS:
Procedure: magnetic resonance imaging. — 1.5 Tesla magnet system is going to be utilized for ankle imaging. A dedicated extremity surface coil (Foot/Ankle 16-Channel Coil; Siemens Medical Solution) is used to enhance spatial resolution.
  Other Names: MRI.

SUMMARY:
Lateral ankle instability may be acute or chronic. Acute instability usually occurs due to extreme rear foot supination with planter-flexion trauma leads to injury of lateral collateral ligament complex especially the anterior talofibular ligament. Most ankle ligamentous injuries are treated conservatively. However, 20% to 40% of patients complain of chronic instability and persistent discomfort. Structural instability, loss of proprioceptive capabilities, and the weakness of peroneal muscles seem to induce chronic instability

ELIGIBILITY:
Inclusion Criteria:

- Patients with any sex, age, complaining of chronic lateral ankle pain.

Exclusion Criteria:

1. Tumors at ankle region.
2. Postoperative status around the ankle.
3. Rheumatoid arthritis.
4. Comminuted fracture at the ankle.
5. Congenital anomalies of the ankle.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with history of ankle trauma or chronic lateral ankle pain that will be evaluated using magnetic resonance imaging.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with ankle or ligaments abnormalities by examination | 30 minutes
  Magnetic resonance imaging examination will be the method for diagnosis